CLINICAL TRIAL: NCT02793024
Title: Shopping Smart - Adolescent Intervention to Improve Shopping Practices Where You Live and Learn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alison Gustafson (Other)
Collaborators: East Carolina University (Other)
Responsible Party: Sponsor-Investigator, Alison Gustafson, Sponsor/Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-0114-PS
Record Dates: First submitted 2016-05-27; First posted 2016-06-08 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Food Choices
Keywords: food shopping intervention
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Intervention (Experimental): Counties will be randomized to receive the intervention or act as a delayed control. Students in the intervention arm will receive the 12-week intervention to improve shopping choices.
  Interventions: Behavioral: Intervention
- Arm 2 - Intervention (No Intervention): Control adolescents will not receive the intervention and will receive routine information normally distributed through schools.

INTERVENTIONS:
Behavioral: Intervention — Adolescents in the intervention arm will receive 3 face to face session about making smart shopping choices. The following 9 weeks will consist of utilizing social media to improve shopping choices.
  Arms: Arm 1 - Intervention

SUMMARY:
The objective of this project is to develop and test the effectiveness of a Cooperative Extension enhanced intervention titled "Smart Shopping," aimed at improving the shopping practices of adolescents with the ultimate goal of increasing fruit and vegetable intake. To achieve this goal, the investigators will conduct formative research (Year 1) via a community-wide analysis of the school, home and neighborhood food environments. In collaboration with Extension staff and faculty, this formative research will provide insight into the development and enhancement of the "Smart Shopping" curriculum (adapted from the "Cooking Matters" Extension curriculum, Year 2). In Years 3-4, the investigators will implement a randomized controlled intervention trial to examine the effectiveness of the developed intervention "Smart Shopping" to improve adolescents' purchasing and consumption behaviors. The investigators will implement the trial in Year 3, and evaluate results in Year 4. Our education component will include training of University dietetics interns, graduate, and undergraduate students to implement and evaluate the intervention with oversight by project staff as part of their service learning requirements. This project is unique as it: 1) takes into account the role that school wellness policies and school environment have in food procurement during the day; 2) incorporates information from multiple levels of the social ecological framework (home, school, and community food environments, as well as the social influence of peers) to create an intervention that addresses influences on adolescents purchasing and consumption behaviors where they live and learn; 3) collaborates with Extension faculty and staff while enhancing an existing program; 4) utilizes and hones the skill sets of students in undergraduate and graduate level nutrition and dietetics programs.

DETAILED DESCRIPTION:
Overview of the study - To achieve sustained healthy behavior changes, a supportive context is needed. For example, adolescents who are trying to consume more fruits and vegetables, fewer sugary beverages, and more water may be challenged in these pursuits as they may be inundated with low-cost, easily available, highly processed foods and beverages. The intervention will take into account the multiple sectors of influence on behavior among adolescents recently recommended. This project moves beyond understanding the interaction between the individual with their environment and seeks to develop and examine the effectiveness of an intervention aiming to improve how adolescents make healthy choices in a variety of food environments and in a variety of social settings.

Overview - This project includes collection of primary data in Year 1 to inform the curriculum development of the "Smart Shopping" intervention in Years 2 and 3. The intervention will take place among 4 schools (2 in KY and 2 in NC) with 4 delayed - control schools (2 in KY and 2 NC). This individual-level intervention will be tailored based on the food environment factors of each site. The key food environmental variables that will be addressed will be school policy adoption and implementation of School Wellness Policies, availability of food within the home, as well as the availability and access to various food venues in each county. After baseline data are collected, the curriculum will be developed reflecting the shopping behaviors of adolescents in these counties. The curriculum will utilize current Cooperative Extension resources from "Cooking Matters," but will be tailored and significantly revised for adolescents using the formative data collected in year 1. The curriculum will be developed with Cooperative Extension agents in each county while connecting with dietetics and nutrition students. The intervention will take place over 12 weeks, once a week, after school but before athletic or school sponsored activities begin. The intervention session will be led by nutrition and dietetics students, with oversight by Cooperative Extension agents and project team. Process evaluation will take place in year 2 and 3 of the study, while main intervention outcome evaluation will take place in year 4 led by project team.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for participation, the adolescent must provide assent and the primary caregiver must provide consent for their child to participate.
* The adolescents must have resided in the county for at least 1 year, plan to reside in the county for at least 1 year, speak English as the primary language, and not report any serious illness that would alter their dietary patterns, such as diabetes or Crohn's disease.
* If there is more than one adolescent in the household within the age range, the adolescent and the primary caregiver will decide which adolescent will participate in the project.

Ages: 14 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
Number of beverage choices per week at baseline and post intervention | 12 weeks
  Beverage intake will be measured with the BEV-Q questionnaire at baseline to determine how many sugar-sweetened beverages and low calories are consumed over a 12 week period among intervention and control participants.
Number of fruit and vegetable servings per week among adolescents at baseline and post intervention | 12 weeks
  Fruit and vegetable serving intake will be measured with the National Cancer Institute Dietary Screener to determine how many servings of fruits and vegetables are consumed over a 12 week period among intervention and control participants.

SECONDARY OUTCOMES:
Availability of fruits and vegetables, water, and sugar-sweetened beverages where adolescents live and shop at baseline and post intervention among intervention and control participants. | 12 weeks
  availability of fruits and vegetables, water, and SSB will be measured through a survey about availability in the home, school, and neighborhood food venues. Questions from Youth Impact and Project EAT survey questions will capture availability.
Frequency of shopping at various food venues baseline and post intervention among intervention and control participants. | 12 weeks
  frequency of shopping at gas stations, convenience stores, and fast-food restaurants compared to controls, as measured by self-report shopping behavior patterns survey7 and key questions from the Youth Impact Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alison Gustafson, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No